CLINICAL TRIAL: NCT05652530
Title: Clinical Study of the Safety and Efficacy of Chimeric Antigen Receptor NK Cell Injection Targeting BCMA (BCMA CAR-NK) in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Clinical Study of the Safety and Efficacy of BCMA CAR-NK
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Pregene Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG2101
Record Dates: First submitted 2022-11-28; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Immunotherapy; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CAR-NK (Experimental)
  Interventions: Drug: Chimeric Antigen Receptor NK Cell Injection Targeting BCMA (BCMA CAR-NK)

INTERVENTIONS:
Drug: Chimeric Antigen Receptor NK Cell Injection Targeting BCMA (BCMA CAR-NK) — This product is allogeneic NK cells which are cryopreserved after in vitro CAR genetic modification and scale-up manufacturing. Subjects are enrolled and treated with lymphocyte clearance chemotherapy (including pre-clearance evaluation), pre-infusion evaluation and BCMA CAR-NK cells infusion.
  Other Names: Lymphocyte clearance

SUMMARY:
The goal of this clinical trial is to study of the Safety and Efficacy of Chimeric Antigen Receptor NK Cell Injection Targeting BCMA (BCMA CAR-NK) in Patients with Relapsed/Refractory Multiple Myeloma

Primary Endpoints:

To evaluate the safety and tolerability of patients with relapsed/refractory multiple myeloma (RR/MM) after BCMA CAR-NK infusion.

To determine the maximum tolerated dose (MTD) and/or subsequent recommended dose (RD) of BCMA CAR-NK in patients with RR/MM.

Secondary Endpoints:

To preliminarily evaluate the effectiveness of BCMA CAR-NK in patients with RR/MM.

To preliminarily evaluate the pharmacokinetic parameters of BCMA CAR-NK cells in patients with RR/MM.

To preliminarily evaluate BCMA CAR-NK cell survival in subjects blood in relation to efficacy, adverse events and relevant biomarker levels.

To preliminarily evaluate the relationship between donors and subjects KIR-Ligand mismatch and safety & efficacy.

To preliminarily evaluate the impact of the degree of HLA genotype matching between donors and subjects on the survival of BCMA CAR-NK cells in the subjects blood.

Subjects are enrolled and treated with lymphocyte clearance chemotherapy (including pre-clearance evaluation), pre-infusion evaluation and BCMA CAR-NK cells infusion and enter the follow-up period after the end of the DLT observation period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above, no gender preference.
* Patients who have received at least 3 prior lines of treatment for multiple myeloma and have failed at least proteasome inhibitor and immunomodulator therapy; Each line has at least 1 complete treatment cycle unless the best remission status for that treatment is documented as progressive disease (PD) (as per the IMWG efficacy evaluation criteria published in 2016, Appendix 4); PD must be documented during or within 12 months after receiving the last treatment.
* Presence of measurable lesions at screening, which are defined as any of the following situations:

Serum M protein≥1 g/dL (≥10 g/L) Urinary M protein≥200 mg/24 hours Serum free light chain (FLC): abnormal serum FLC ratio (<0.26 or >1.65) and involved FLC≥10 mg/dL (100 mg/L)

* ECOG score (Appendix 1): 0~1.
* Expected survival≥3 months.
* The following test values within 7 days prior to lymphocyte clearance meet the following criteria:

Hematology Absolute lymphocyte count:≥0.5×109/L[Granulocyte colony-stimulating factor (G-CSF) is allowed, but subjects should not have received this supportive therapy within 7 days prior to laboratory test during the screening period] Absolute neutrophil count:≥1.0×10^9 /L[Granulocyte colony-stimulating factor (G-CSF) is allowed, but subjects should not have received this supportive therapy within 7 days prior to laboratory test during the screening period].

Platelets:Subjects platelet count ≥50 x 10^9/L (subjects must not receive transfusion support within 7 days prior to laboratory test during the screening period) Hemoglobin:≥8.0 g/dL (recombinant human erythropoietin is allowed) [subjects have not received a red blood cell (RBC) transfusion within 7 days prior to laboratory test during the screening period].

Liver Total bilirubin (serum) :Total bilirubin (serum) ≤1.5 × ULN AST and ALT:≤3× ULN

* Peripheral venous pathway meets the requirements of intravenous drip.
* Subjects agree to use reliable methods for contraception from the time of signing the informed consent till 1 year after the transfusion.
* Voluntary participation in the clinical trial and signing of the informed consent form.

Exclusion Criteria:

* Subjects who have had a severe anaphylactic reaction.
* Subjects who received the following anti-MM therapy within a specific time prior to lymphocyte clearance.

Small molecule targeted therapy within 2 weeks or 5 half-lives (whichever is longer).

Large-molecule drug within 4 weeks or 2 half-lives (whichever is longer). Cytotoxic drugs, modern Chinese medicine preparations with antitumor effects within 2 weeks.

Immunomodulators therapy within 1 week.

* Subjects who have received a live or attenuated vaccine within 4 weeks prior to lymphocyte clearance.
* Subjects who have received the following therapy within 7 days prior to lymphocyte clearance, or that requires long-term treatment during the study period according to the investigators:

Systemic steroid therapy (except for inhaled one or topical use). Immunosuppressive therapy. Treatment of graft-versus-host response.

* Subjects presenting with incomplete recovery or stabilization to grade 1 (NCI-CTCAE v5.0) of toxicity (including peripheral neuropathy) caused by prior treatments.
* Cardiac disease: episode of myocardial infarction≤6 months prior to lymphocyte clearance; episode of unstable angina, severe arrhythmia as judged by the investigators, or coronary artery bypass graft≤3 months prior to lymphocyte clearance.
* Women who are pregnant or breastfeeding.
* Subjects who, in the opinion of the investigators, have any clinical or laboratory test abnormalities or other reasons that make them ineligible to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-11-13 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Toxicity Assessment per Adverse Event reporting classified according to CTCAE V5.0 | Day 28
  per Adverse Event reporting classified according to CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No